CLINICAL TRIAL: NCT04646824
Title: A Study of Almonertinib With Chemotherapy as 1st Line Treatment in Patients With Mutated Epidermal Growth Factor Receptor Non-Small Cell Lung Cancer
Brief Title: Almonertinib With Chemotherapy in mEGFR NSCLC
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Tianjin Medical University Cancer Institute and Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ahead001
Record Dates: First submitted 2020-11-19; First posted 2020-11-30 (Actual); Last update posted 2020-12-02 (Actual); Status verified 2020-11

CONDITIONS: Non-Small Cell Lung Cancer Metastatic
MeSH Terms: interventions — Cisplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- ahead (Experimental): A110 mg QD and platinum-based chemotherapy. A 110 mg in combination with pemetrexed (500 mg/m2) plus cisplatin (75 mg/m2) or carboplatin (AUC5) on Day 1 of 21day cycles (every 3 weeks) for 4 cycles, followed by A 110mg daily with pemetrexed maintenance (500 mg/m2) every 3 weeks. Dose may be reduced to allow for the management of IP related toxicity.
  Interventions: Drug: Almonertinib Pemetrexed/Cisplatin

INTERVENTIONS:
Drug: Almonertinib Pemetrexed/Cisplatin — Pemetrexed/Cisplatin Drug: Pemetrexed (500 mg/m2) plus cisplatin (75 mg/m2) on Day 1 of 21day cycles (every 3 weeks) for 4 cycles, followed by Almonertinib daily with pemetrexed maintenance (500 mg/m2) every 3 weeks.

SUMMARY:
The reason for the study is to find out if an experimental combination of an oral medication called Almonertinib when used in combination with chemotherapy is more effective for the treatment of locally advanced or metastatic non-small cell lung cancer. Some lung cancers are due to mutations in the Deoxyribonucleic acid (DNA) which, if known, can help physicians decide the best treatment for patients. One type of mutation can occur in the gene that produces a protein on the surface of cells called the Epidermal Growth Factor Receptor (EGFR).

DETAILED DESCRIPTION:
In total the study aims to enroll approximately 36 patients who will receive almonertinib in combination with chemotherapy in the main trial. The study involves a Screening Period, Treatment Period, and Follow up Period. Whilst receiving study medication, it is expected patients will attend, on average, approximately 15 visits over the first 12 months and then approximately 4 visits per year afterwards. Each visit will last about 2 to 6 hours depending on the arrangement of medical assessments by the study centre.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female, at least 18 years of age; patients from Japan at least 20 years of age.
2. Pathologically confirmed non-squamous Non-Small Cell Lung Cancer (NSCLC).
3. Newly diagnosed locally advanced (clinical stage IIIB, IIIC) or metastatic Non-Small Cell Lung Cancer (NSCLC) (clinical stage IVA or IVB) or recurrent Non-Small Cell Lung Cancer (NSCLC) not amenable to curative surgery or radiotherapy.
4. The tumor harbors 1 of the 2 common epidermal growth factor receptor (EGFR) mutations known to be associated with Epidermal growth factor receptor tyrosine kinase inhibitors (EGFR-TKI) sensitivity (Ex19del or L858R), either alone or in combination with other epidermal growth factor receptor (EGFR) mutations, which may include T790M.
5. Patients must have untreated advanced Non-Small Cell Lung Cancer (NSCLC) not amenable to curative surgery or radiotherapy.
6. WHO PS of 0 to 1 at screening with no clinically significant deterioration in the previous 2 weeks.
7. Life expectancy >12 weeks at Day 1.
8. Willing to use contraception as appropriate during the study and for a period of time after discontinuing study treatment.

Exclusion Criteria:

1. Spinal cord compression; symptomatic and unstable brain metastases, except for those patients who have completed definitive therapy, are not on steroids, and have a stable neurological status for at least 2 weeks after completion of the definitive therapy and steroids.
2. Past medical history of Interstitial Lung Disease (ILD), drug-induced Interstitial Lung Disease, radiation pneumonitis that required steroid treatment, or any evidence of clinically active Interstitial Lung Disease.
3. Any evidence of severe or uncontrolled systemic diseases, including uncontrolled hypertension and active bleeding diatheses, which in the Investigator's opinion makes it undesirable for the patient to participate in the trial.
4. QT prolongation or any clinically important abnormalities in rhythm.
5. Inadequate bone marrow reserve or organ function as demonstrated by any of the following laboratory values:
6. Refractory nausea and vomiting, chronic gastrointestinal diseases, inability to swallow the formulated product, or previous significant bowel resection that would preclude adequate absorption of osimertinib.
7. Prior treatment with any systemic anti-cancer therapy for advanced Non-Small Cell Lung Cancer (NSCLC) not amenable to curative surgery or radiation including chemotherapy, biologic therapy, immunotherapy, or any investigational drug. Prior adjuvant and neo-adjuvant therapies (chemotherapy, radiotherapy, immunotherapy, biologic therapy, investigational agents), or definitive radiation/chemoradiation with or without regimens including immunotherapy, biologic therapies, investigational agents are permitted as long as treatment was completed at least 12 months prior to the development of recurrent disease.
8. Prior treatment with an Epidermal growth factor receptor tyrosine kinase inhibitors (EGFR-TKI).
9. Major surgery within 4 weeks of the first dose of investigational product (IP). Procedures such as placement of vascular access, biopsy via mediastinoscopy or biopsy via video assisted thoracoscopic surgery are permitted.
10. Radiotherapy treatment to more than 30% of the bone marrow or( with a wide field of radiation within 4 weeks of the first dose of investigational product (IP). -
11. History of hypersensitivity to active or inactive excipients of investigational product (IP) or drugs with a similar chemical structure or class to investigational product (IP)

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2020-11-19 (Actual); Primary Completion 2020-11-28 (Estimated); Study Completion 2022-11-25 (Estimated)

PRIMARY OUTCOMES:
PFS | The primary analysis of Progressionfree survival (PFS) based on investigator assessment will occur when PFS maturity is observed at approximately 33 months
  Progression-free survival

CONTACTS AND LOCATIONS:
Locations (1):
- Tianjin Medical University Cancer Institute and Hospital, Tianjin, Tianjin Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided